CLINICAL TRIAL: NCT00489203
Title: A Phase II Study to Evaluate the Efficacy of Oral Beclomethasone Dipropionate for Prevention of Acute GVHD After Hematopoietic Cell Transplantation With Myeloablative Conditioning Regimens
Brief Title: Beclomethasone Dipropionate in Preventing Acute Graft-Versus-Host Disease in Patients Undergoing a Donor Stem Cell Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2079.00; NCI-2009-01544
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2015-03

CONDITIONS: Hematopoietic/Lymphoid Cancer; Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; de Novo Myelodysplastic Syndromes; Essential Thrombocythemia; Extramedullary Plasmacytoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Graft Versus Host Disease; Isolated Plasmacytoma of Bone; Juvenile Myelomonocytic Leukemia; Meningeal Chronic Myelogenous Leukemia; Myelodysplastic/Myeloproliferative Disease, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Childhood Hodgkin Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage I Mycosis Fungoides/Sezary Syndrome; Stage I Small Lymphocytic Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Multiple Myeloma; Stage II Mycosis Fungoides/Sezary Syndrome; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Thrombocythemia, Essential; Graft vs Host Disease; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Lymphoma, Large-Cell, Immunoblastic; Multiple Myeloma | interventions — Beclomethasone; Tacrolimus; Methotrexate; merphos

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral beclomethasone dipropionate 4 times daily beginning at the start of the conditioning regimen and continuing through day 75 post-transplant. Patients also receive a standard immunosuppressive regimen comprising tacrolimus and methotrexate post-transplant.
  Interventions: Drug: beclomethasone dipropionate; Drug: tacrolimus; Drug: methotrexate; Procedure: allogeneic hematopoietic stem cell transplantation
- Arm II (Active Comparator): Patients receive oral placebo 4 times daily beginning at the start of the conditioning regimen and continuing through day 75 post-transplant. Patients also receive a standard immunosuppressive regimen comprising tacrolimus and methotrexate post-transplant.
  Interventions: Drug: placebo; Drug: tacrolimus; Drug: methotrexate; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: beclomethasone dipropionate — Given orally
  Other Names: BECLOMETH; Beclovent; Beconase; Qvar; Vancenase; Vanceril
  Arms: Arm I
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II
Drug: tacrolimus — Given after transplant
  Other Names: Advagraf; FK 506; Prograf; Protopic
Drug: methotrexate — Given after transplant
  Other Names: Abitrexate; amethopterin; Folex; methylaminopterin; Mexate; MTX
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo stem cell transplant

SUMMARY:
RATIONALE: Beclomethasone dipropionate may be effective in preventing acute graft-versus-host disease in patients undergoing a stem cell transplant for hematologic cancer.

PURPOSE: This randomized phase II trial is studying how well beclomethasone dipropionate works in preventing acute graft-versus-host disease in patients undergoing a donor stem cell transplant for hematologic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the efficacy of oral BDP for prevention of acute GVHD after allogeneic hematopoietic cell transplantation with myeloablative conditioning regimens.

OUTLINE:

Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral beclomethasone dipropionate 4 times daily beginning at the start of the conditioning regimen and continuing through day 75 post-transplant. Patients also receive a standard immunosuppressive regimen comprising tacrolimus and methotrexate post-transplant.

ARM II: Patients receive oral placebo 4 times daily beginning at the start of the conditioning regimen and continuing through day 75 post-transplant. Patients also receive a standard immunosuppressive regimen comprising tacrolimus and methotrexate post-transplant.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion

* Allogeneic HCT with marrow or growth-factor mobilized blood cells from an HLA-A, B, C, DRB1, and HLA-DQB1-allele matched or single-allele or antigen mismatched related or unrelated donor
* Use of myeloablative pre-transplant conditioning regimen with > 800 cGy total body irradiation and cyclophosphamide, or high-dose busulfan and cyclophosphamide
* Use of methotrexate and tacrolimus for prevention of GVHD after allogeneic HCT
* Informed consent document signed

Exclusion

* Cord blood transplant recipients
* Use of T cell depletion or rabbit antithymocyte globulin to prevent acute GVHD
* Treatment with rabbit antithymocyte globulin or alemtuzumab within 3 months before the date of HCT
* Participation in another therapeutic trial where the primary endpoint is related to acute GVHD
* Hospitalization at the beginning of the pre-transplant conditioning regimen because of pre-existing medical complications
* Glucocorticoid treatment at prednisone-equivalent doses > 0.2 mg/kg/day
* Known intolerance to BDP
* Anticipated inability to tolerate oral administration of study drug tablets for any reason during the first two weeks after HCT
* Body weight < 35 kg (lower-dose formulations are not available for subjects with lower body weight)
* Pregnancy or breast feeding
* Women of child-bearing potential who are unwilling to use a reliable method of contraception
* Incarceration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-04; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Development of acute graft-versus-host disease (GVHD) with severity sufficient to require systemic immunosuppressive treatment | On or before day 90 after the transplant

SECONDARY OUTCOMES:
Cumulative glucocorticoid dose (measured as prednisone equivalents) per kg body weight | First 75 days after HCT
Peak and average skin, liver and gut morbidity stages and overall grades | To day 90 after HCT
Modified average acute GVHD index score | To day 90 after HCT
Cumulative incidence of systemic immunosuppressive treatment for acute GVHD | At any time after HCT
Cumulative incidence of topical therapy for acute GVHD, including psoralen and UV irradiation, hydrocortisone cream, topical tacrolimus, oral BDP, or oral swish and spit dexamethasone | On or before day 90 after the transplant
Cumulative incidence of biopsy-proven gastrointestinal GVHD | On or before day 90 after the transplant
Proportion of patients with grade IIa GVHD | On or before day 90 after the transplant
Proportions of patients with grades IIa and IIb - IV GVHD | On or before day 90 after the transplant
Cumulative incidence of chronic GVHD requiring systemic immunosuppressive treatment | At any time after HCT
Number of days in the hospital | During the first 90 days after HCT
Non-relapse mortality | At any time after HCT
Overall survival | At any time after HCT
Survival | At 200 days after HCT
Safety | On or before day 90 after the transplant
Feasibility | First 75 days after HCT
Survival without recurrent malignancy | At any time after HCT

CONTACTS AND LOCATIONS:
Overall Officials: Paul Martin, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Fred Hutchinson Cancer Research Center, Seattle, Washington